CLINICAL TRIAL: NCT01878526
Title: The Effectiveness of Domperidone Versus Alginic Acid Add on Omeprazole Therapy in Omeprazole Resistance Gastroesophageal Reflux in Systemic Sclerosis
Brief Title: Gastroesophageal Reflux Treatment in Scleroderma
Acronym: GERD-SSc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Chingching Foocharoen, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GERD therapy in scleroderma; PPI in SSc-GERD (Other Grant/Funding Number: Thai Rheumatism Association)
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Gastroesophageal Reflux Disease; Systemic Sclerosis; Scleroderma
Keywords: gastroesophageal reflux disease; heart burn; regurgitation; systemic sclerosis; scleroderma; proton pump inhibitor; alginic acid; omeprazole; prokinetic
MeSH Terms: conditions — Gastroesophageal Reflux; Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Alginic Acid; Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omeprazole plus alginic acid and placebo of domperidone (Experimental)
  Interventions: Drug: Alginic acid; Drug: placebo (for domperidone)
- Omeprazole plus domperidone and placebo of alginic acid (Experimental)
  Interventions: Drug: Domperidone; Drug: placebo (of alginic acid)

INTERVENTIONS:
Drug: Alginic acid — Algycon 1 tab chew tid after meal
  Other Names: Algycon
  Arms: Omeprazole plus alginic acid and placebo of domperidone
Drug: placebo (for domperidone) — placebo (for domperidone) 1 tab oral tid before meal
  Arms: Omeprazole plus alginic acid and placebo of domperidone
Drug: Domperidone — domperidone (10 mg) 1 tab oral tid before meal
  Other Names: Molax
  Arms: Omeprazole plus domperidone and placebo of alginic acid
Drug: placebo (of alginic acid) — placebo (for alginic acid) 1 tab chew tid after meal
  Arms: Omeprazole plus domperidone and placebo of alginic acid

SUMMARY:
The investigators purposes are to define the prevalence of omeprazole resistance gastroesophageal reflux disease (GERD) in systemic sclerosis (SSc), to compare the efficacy of omeprazole in combination with algycon versus omeprazole in combination with domperidone on the severity of reflux symptoms in omeprazole resistant GERD in SSc, and to compare the efficacy of omeprazole in combination with algycon versus omeprazole in combination with domperidone on the frequency of symptoms in omeprazole- resistant GERD in SSc.

ELIGIBILITY:
Phase 1 SSc patients who fit all inclusion and exclusion criteria will be eligible to phase 1 study for evaluation the prevalence of omeprazole resistant-GERD

Inclusion criteria:

1. SSc patients aged between 18 and 65 years.
2. Clinically diagnosed as GERD and GERD-questionnaire score >3
3. Must not receive any proton pump inhibitor (PPI) or prokinetic drug within 2 weeks before baseline evaluation

Exclusion criteria:

1. Pregnancy or lactation
2. Previous history of gastroesophageal surgery or endoscopic therapy due to severe erosive esophagitis
3. Present of Barrett's esophagus
4. Bedridden and confined to no self-care
5. Evidence of active malignant disease
6. Present of uncontrolled or severe medical problems such as asthma, angina, hepatic or renal diseases
7. Present of active infection that needs systemic antibiotic
8. Allergic history of omeprazole
9. Receiving prohibit co-medications that may have drug interaction or attenuate GERD symptoms such as tetracycline, ferrous salt, digoxin, isoniacid, oral bisphosphonate

Phase 2 randomized parallel study SSc patients who fit all inclusion and exclusion criteria will be eligible to phase 2 study.

Inclusion criteria:

1. SSc patients who completed the phase 1 study.
2. The subjects were defined as PPI-resistance.
3. The subject must be willing to continue phase 2 study.

Exclusion criteria:

1. Pregnancy
2. Present of uncontrolled or severe medical problems
3. Present of active infection
4. Allergic history of alginic acid or domperidone
5. Receiving prohibit co-medications that may have drug interaction or attenuate GERD symptoms such as tetracycline, ferrous salt, digoxin, isoniacid, oral bisphosphonate
6. Chewing difficulty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chingching Foocharoen, MD, Principal Investigator — Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- 123 Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Foocharoen C, Chunlertrith K, Mairiang P, Mahakkanukrauh A, Suwannaroj S, Namvijit S, Wantha O, Nanagara R. Effectiveness of add-on therapy with domperidone vs alginic acid in proton pump inhibitor partial response gastro-oesophageal reflux disease in systemic sclerosis: randomized placebo-controlled trial. Rheumatology (Oxford). 2017 Feb;56(2):214-222. doi: 10.1093/rheumatology/kew216. Epub 2016 May 13. PMID 27179107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Started | 40 | 40
Completed | 37 | 38
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (9.5) | 46.7 (12.5) | 48.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 30 | 47
  Male | 20 | 8 | 28
Region of Enrollment [Number; unit: participants]
  Thailand | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Changing Severity of Heart Burn of SSc Related Omeprazole Resistant GERD Evaluated by Visual Analogue Score (VAS)
Description: VAS scale 0-100 was applied for an outcome measurement of the severity of heart burn. The VAS scale 0 was no symptoms of heart burn and scale 100 was a maximum symptom of heart burn. The changing of the severity of heart burn was the changing of VAS before and after treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: VAS (100)
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Number analyzed (Participants) | 37 | 38
VAS (100) | 17.9 (13.1) | 17.2 (13.9)

2. Primary Outcome: Changing of the Severity of Regurgitation
Description: VAS scale 0-100 was applied for an outcome measurement of the severity of regurgitation. The VAS scale 0 was no symptoms of regurgitation and scale 100 was a maximum symptom of regurgitation. The changing of the severity of regurgitation was the changing of VAS before and after treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: VAS (100)
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Number analyzed (Participants) | 37 | 38
VAS (100) | 24.9 (15.9) | 23.1 (15.1)

3. Secondary Outcome: Changing of Frequency of Symptoms in SSc Related Omeprazole Resistant GERD Evaluated by Frequency Scale for the Symptoms of GERD (FSSG)
Description: Unit scale 0-48 was applied for an outcome measurement of the frequency of symptoms. The unit scale 0 was no symptom and scale 48 was usual symptom of GERD. The changing of the frequency of symptoms was the changing of the unit scale before and after treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Number analyzed (Participants) | 37 | 38
units on a scale | 4.6 (3.3) | 4.7 (3.7)

4. Secondary Outcome: the Prevalence of Omeprazole-resistant GERD in SSc After 4 Weeks Treatment With Omeprazole
Time Frame: 4 weeks
Population: The number of analysed patients came out the total number of screening patients in the trial. The patients who were defined as omeprazole-resistant GERD were enrolled and randomized for either alginic acid plus placebo or domperidone plus placebo group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall Systemic Sclerosis With GERD (Before Randomization): omeprazole 20 mg bid ac for 4 weeks for overall systemic sclerosis with GERD
Arm/Group | Overall Systemic Sclerosis With GERD (Before Randomization)
Number analyzed (Participants) | 148
percentage of participants | 59 [51 to 67]

5. Secondary Outcome: Changing of the Quality of Life Which is Evaluated by EQ-5DTM
Description: VAS scale 0-100 was applied for an outcome measurement of the quality of life. The VAS scale 0 was the worst quality of life and scale 100 was the best quality of life. The changing of the quality of life was the changing of VAS of quality of life before and after treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: VAS (100)
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Number analyzed (Participants) | 37 | 38
VAS (100) | 75.7 (15.8) | 76.1 (14.4)

ADVERSE EVENTS:
Arm/Group | Omeprazole Plus Alginic Acid and Placebo of Domperidone | Omeprazole Plus Domperidone and Placebo of Alginic Acid
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 2/37 | 2/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omeprazole Plus Alginic Acid and Placebo of Domperidone (N=37) | Omeprazole Plus Domperidone and Placebo of Alginic Acid (N=38)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No